CLINICAL TRIAL: NCT01360814
Title: A Structured Multidisciplinary Intervention to Improve Quality of Life of Patients Receiving Active Oncological Treatment: A Randomized Trial
Brief Title: Structured Multidisciplinary Intervention or Standard Medical Care in Improving Quality of Life in Patients Receiving Active Cancer Treatment
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC0491; NCI-2011-00670 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC0491 (Other: Mayo Clinic Cancer Center); 2314-04 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2011-05-23; First posted 2011-05-26 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-05

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Counseling; Early Intervention, Educational; Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- GROUP A (multidisciplinary intervention): Patients receive six 90-minute sessions of a multidisciplinary structured intervention comprising physical therapy, education, a cognitive-behavioral intervention, discussion and support, spiritual reflection, and a relaxation exercise over 2-4 weeks. Caregivers are invited to sessions 1, 3, 4, and 6. Patients may also receive brief telephone contact during the 6 month follow-up period.
  Interventions: Procedure: quality-of-life assessment; Behavioral: telephone-based intervention; Other: questionnaire administration; Other: counseling intervention; Behavioral: exercise intervention; Other: educational intervention
- GROUP B (standard medical care): Patients receive standard medical care only. Patients may also receive brief telephone contact during the 6 month follow-up period.
  Interventions: Procedure: quality-of-life assessment; Other: questionnaire administration; Behavioral: telephone-based intervention; Procedure: standard follow-up care

INTERVENTIONS:
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Behavioral: telephone-based intervention — Receive multidisciplinary structured intervention
  Groups: GROUP A (multidisciplinary intervention)
Other: questionnaire administration — Ancillary studies
Other: counseling intervention — Receive multidisciplinary structured intervention
  Other Names: counseling and communications studies
  Groups: GROUP A (multidisciplinary intervention)
Behavioral: exercise intervention — Receive multidisciplinary structured intervention
  Groups: GROUP A (multidisciplinary intervention)
Other: educational intervention — Receive multidisciplinary structured intervention
  Other Names: intervention, educational
  Groups: GROUP A (multidisciplinary intervention)
Behavioral: telephone-based intervention — Receive standard care
  Groups: GROUP B (standard medical care)
Procedure: standard follow-up care — Receive standard care
  Groups: GROUP B (standard medical care)

SUMMARY:
This randomized clinical trial studies structured multidisciplinary intervention or standard medical care in improving quality of life (QOL) in patients receiving active cancer treatment. A structured multidisciplinary intervention may improve the QOL in patients receiving treatment for cancer. It is not yet known whether structured multidisciplinary intervention is more effective than standard medical care in improving QOL

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the efficacy of a structured multidisciplinary intervention compared to standard medical care on improving the subject's QOL as measured by the Functional Assessment of Cancer Therapy-General global summary score (FACT-G) at 4 weeks (or at end of the intervention), at 27 weeks and at 52 weeks.

SECONDARY OBJECTIVES:

I. To examine the effect of a structured multidisciplinary intervention compared to standard medical care on improving the subject's psychosocial functioning as measured by the 11 Linear Analogue Self Assessment (LASA) QOL scales, Profile of Mood States (POMS), the Functional Assessment of Chronic Illness Therapy-Spiritual well-being scale (FACIT-SP), Pittsburgh Sleep Quality Index, the Epworth Sleepiness Scale, the Control Preferences Scale, and Exercise Behaviors at 4 weeks (or at end of intervention), at 27 weeks and at 52 weeks.

II. To examine the effect of a structured multidisciplinary intervention compared to standard medical care on improving the caregiver's QOL as measured by the Caregiver QOL-Cancer scale, and on their psychosocial functioning as measured by the 11 LASA QOL scales and POMS at 4, 27 and 52 weeks.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP A: Patients receive six 90-minute sessions of multidisciplinary structured intervention comprising physical therapy, education, a cognitive-behavioral intervention, discussion and support, spiritual reflection, and a relaxation exercise over 2-4 weeks. Caregivers are invited to sessions 1, 3, 4, and 6. Patients may also receive brief telephone contact during the 6 month follow-up period.

GROUP B: Patients receive standard medical care only. Patients may also receive brief telephone contact during the 6 month follow-up period.

After completion of study treatment, patients are followed up at 4 weeks (or at the end of intervention), at 27 weeks, and at 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ability to attend all treatment sessions and follow-up
* Ability to provide written informed consent
* Ability to participate in all aspects of the study
* Initial diagnosis of cancer must have been =< 12 months prior to study entry
* Intermediate to poor prognosis, defined as an expected 5-year survival of 0-50% in the judgment of the physicians entering the patient on the study
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1, or 2
* >= 1 week of planned cancer treatment at Mayo Clinic
* Has a caregiver also willing to participate

Exclusion Criteria:

* Mini-mental state examination (MMSE) scores of < 20
* Expected survival of < 6 months
* Active substance abuse (alcohol or drug)
* Participation in other psycho-social research trials
* Active thought disorder (bipolar illness, schizophrenia, etc.)
* Suicidal intent or plan
* In need of psychiatric hospitalization
* Recurrent disease after disease-free interval of > 6 months
* Previous cancer =< 5 years (except non-melanoma skin cancer and/or second cancer diagnosed at approximately the same time as this cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2009-03-13 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Cancer patient's quality of life (QOL) as measured by the FACT-G global summary score | At baseline and 4, 27, and 52 weeks
  The t-test and Wilcoxon test supplemented by repeated measures analytical procedures (analysis of variance [ANOVA], Generalized Estimating Equations [GEE]) will be used to measure and analyze QOL.

SECONDARY OUTCOMES:
On improving the subject's psychosocial functioning as measured by the 11 LASA QOL scales, Profile of Mood States (POMS), the FACIT-SP, Pittsburgh Sleep Quality Index, the Epworth Sleepiness Scale, the Control Preferences Scale, and Exercise Behaviors | At baseline and 4, 27, and 52 weeks
  The t-test and Wilcoxon test supplemented by repeated measures analytical procedures (analysis of variance [ANOVA], Generalized Estimating Equations [GEE]) will be used to measure and analyze.
On improving the caregiver's QOL as measured by the Caregiver QOLCancer scale, and on their psychosocial functioning as measured by the 11 LASA QOL scales and POMS | At baseline and 4, 27 and 52 weeks
  The t-test and Wilcoxon test supplemented by repeated measures analytical procedures (analysis of variance [ANOVA], Generalized Estimating Equations [GEE]) will be used to measure and analyze

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Clark, Ph.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Chock MM, Lapid MI, Atherton PJ, Kung S, Sloan JA, Richardson JW, Clark MM, Rummans TA. Impact of a structured multidisciplinary intervention on quality of life of older adults with advanced cancer. Int Psychogeriatr. 2013 Dec;25(12):2077-86. doi: 10.1017/S1041610213001452. Epub 2013 Sep 4. PMID 24001635